CLINICAL TRIAL: NCT01106716
Title: A Double-Blind, Randomized, Placebo- and Active-Comparator-Controlled, Single-Dose Study to Assess the Efficacy of KAI-1678 Administered by Subcutaneous Infusion in Subjects With Postherpetic Neuralgia
Brief Title: Safety and Efficacy Study of KAI-1678 to Treat Pain in Subjects With Postherpetic Neuralgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KAI Pharmaceuticals (Industry)
Collaborators: Trident Clinical Research Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KAI-1678-003
Record Dates: First submitted 2010-04-16; First posted 2010-04-20 (Estimated); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Postherpetic Neuralgia
Keywords: Lidocaine; Lignocaine; Analgesics. Non-narcotic / therapeutic use; Neuralgia, Postherpetic; Pain; Pain measurement / drug effect; Pain postoperative / drug therapy; PHN
MeSH Terms: conditions — Neuralgia, Postherpetic; Pain; Pain, Postoperative | interventions — KAI-1678; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A1: Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- A2: KAI-1678 (Experimental): Experimental
  Interventions: Drug: KAI-1678
- A3: Lidocaine (Active Comparator): Lidocaine
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Placebo — Placebo IV Infusion
  Arms: A1: Placebo
Drug: KAI-1678 — KAI-1678 IV Infusion
  Arms: A2: KAI-1678
Drug: Lidocaine — Lidocaine
  Arms: A3: Lidocaine

SUMMARY:
The purpose of this study is to determine whether KAI-1678 is effective in the treatment of postherpetic neuralgia pain

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PHN with pain for at least 3 months after segmental herpes zoster eruption
* pain score at least 4 on 11-point numerical rating scale (0-10)
* stable doses of analgesic medications for at least 1 month"

Exclusion Criteria:

* diagnosis of PHN with pain for at least 3 months after segmental herpes zoster eruption
* pain score at least 4 on 11-point numerical rating scale (0-10)
* stable doses of analgesic medications for at least 1 month"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The effect of KAI-1678 on mean change from baseline in pain intensity at 6 hours (PID 6). | Day 1
  Measurements are made using a qualified pain scale and the change from basline is calculated at 6 hours.

SECONDARY OUTCOMES:
The effect of KAI-1678 on the proportion of subjects achieving at least a 1 point improvement in pain intensity at 6 hours | Day 1
The effect of KAI-1678 on patient global response to treatment | Day 1
The effect of KAI-1678 on symptoms associated with PHN assessed by the Neuropathic Pain Scale (NPS) | Day 1
The number of adverse events as a measure of safety and tolerability of KAI-1678 | Two weeks
  Frequency of adverse events on each study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Bell, MD, Study Director — KAI Pharmaceuticals, Inc
Locations (1):
- Sydney, New South Wales, Australia